CLINICAL TRIAL: NCT04820491
Title: EASiUR Trial: Efficient Anterior Shoulder Ultrasound Reduction Multicenter Prospective Randomized Trial
Brief Title: Efficient Anterior Shoulder Ultrasound Reduction Multicenter Prospective Randomized Trial
Acronym: EASiUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HM20019991
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation | interventions — X-Rays; Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- X-Ray (Active Comparator)
  Interventions: Diagnostic Test: X-Ray
- Ultrasound (Active Comparator)
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: X-Ray — Shoulder x-rays as felt necessary for standard of care of diagnosis of shoulder dislocation and reduction
  Arms: X-Ray
Diagnostic Test: Ultrasound — Initial evaluation with ultrasound; may also evaluate nearby areas for concern of fracture. Order x- rays after ultrasound as seen fit for other injuries of diagnostic uncertainty.
  Arms: Ultrasound

SUMMARY:
The purpose of the study is to determine if using ultrasound to diagnosis and confirm reductions of shoulder dislocations impacts the length of an emergency department visit for this condition.

DETAILED DESCRIPTION:
The purpose of the study is to determine if the length of the emergency department visit can be decreased and if patient exposure to x-rays can be reduced by utilizing an ultrasound to diagnose and confirm reduction in shoulder dislocations.

This study also seeks to determine if patients prefer ultrasound to x-ray when used to treat their shoulder dislocation.

Participants will be randomly assigned to one of two groups: either x-rays or ultrasound for the diagnosis and reduction confirmation of your shoulder dislocation.

Participant's shoulder dislocation will be treated per standard of care.

Participants will be asked to complete a short survey at the end of their visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years of age or older; and
2. Present to the VCU Emergency Department; and
3. Have clinical signs of uncomplicated shoulder dislocation; and
4. Agree to participation in the study; and
5. Provides a written consent to be included in the study.

Exclusion Criteria:

1. Patients who have a level 1 or 2 trauma activation, and/or;
2. Patients who are pregnant, incarcerated, or unable to consent, and/or;
3. Patients who have a past medical history of shoulder replacement in dislocated shoulder; and/or
4. Provider Discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Tozer, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | X-Ray | Ultrasound
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data was not collected directly from participants but was to be extracted from participant charts. Data was not extracted from patient charts due to termination of the study and in compliance with the HIPAA "Minimum Necessary" standard.
Groups:
- Total: Total of all reporting groups
Arm/Group | X-Ray | Ultrasound | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Customized [Number; unit: participants] — Demographic data was not collected directly from participants but was to be extracted from participant charts. Data was not extracted from patient charts due to termination of the study and in compliance with the HIPAA "Minimum Necessary" standard.
  participants
    Unknown | 5 | 4 | 9
Sex/Gender, Customized [Count of Participants; unit: Participants] — Demographic data was not collected directly from participants but was to be extracted from participant charts. Data was not extracted from patient charts due to termination of the study and in compliance with the HIPAA "Minimum Necessary" standard.
  Participants
    Unknown | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay in the Emergency Department (ED)
Description: Length of stay in the ED will be calculated from time of first provider contact to time of discharge from the ED.
Time Frame: up to 8 hours or time to admission
Population: Data was not extracted from patient charts due to termination of the study and in compliance with the HIPAA "Minimum Necessary" standard.
Arm/Group | X-Ray | Ultrasound
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction will be assessed using a 6 item scale. Each item is rated from 1 (extremely dissatisfied) to 5 (extremely satisfied). Scores are summed yielding scores ranging from 6 (most dissatisfied) to 30 (most satisfied).
Time Frame: at discharge or admission - up to 8 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | X-Ray | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 29.25 (0.96) | 27.75 (2.06)

3. Secondary Outcome: Time to Diagnosis
Description: Time to diagnosis will be calculated from time of first provider contact to time of x-ray or time of ultrasound per treatment condition
Time Frame: up to 8 hours or time to admission
Population: as for outcome 1
Arm/Group | X-Ray | Ultrasound
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Confirmation of Reduction
Description: As documented by x-ray or ultrasound per treatment condition
Time Frame: up to 8 hours or time to admission
Population: as for outcome 1
Arm/Group | X-Ray | Ultrasound
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cost of Treatment
Description: Calculated as total billing cost of procedures related to shoulder dislocation ED visit
Time Frame: up to 8 hours or time to admission
Population: as for outcome 1
Arm/Group | X-Ray | Ultrasound
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Total Number of Xrays
Description: Total number of xrays ordered during time in ED
Time Frame: up to 8 hours or time to admission
Population: as for outcome 1
Arm/Group | X-Ray | Ultrasound
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 hours
Arm/Group | X-Ray | Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04820491/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04820491/ICF_001.pdf